CLINICAL TRIAL: NCT04669132
Title: Efficacy of Olanzapine, Netupitant and Palonosetron in Controlling Nausea and Vomiting Associated With Highly Emetogenic Chemotherapy in Patients With Breast Cancer
Acronym: OLNEPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Camilla Vieira de Rebouças, MD, Instituto Brasileiro de Controle do Cancer
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38285020.8.0000.0072
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Nausea Post Chemotherapy
Keywords: olanzapine; emetogenic; chemotherapy; breast cancer; nausea
MeSH Terms: conditions — Breast Neoplasms; Nausea | interventions — Olanzapine; netupitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olanzapine + Netupitanto + Palonosetron (Experimental): Olanzapine 5 mg/day d 0-4 + Netupitanto 300 mg/day d 1 + Palonosetron 0.56 mg/day d 1;
  Interventions: Drug: Olanzapine; Drug: Netupitant; Drug: Palonesetron

INTERVENTIONS:
Drug: Olanzapine — - Olanzapine 5mg, administered once daily, during 5 days (day before chemotherapy, the D day of the chemotherapy and 3 day after chemotherapy)
Drug: Netupitant — - Netupitanto 300 mg, once daily, on chemotherapy day;
Drug: Palonesetron — - Palonosetron 0.56 mg, once daily, on chemotherapy day;

SUMMARY:
This is a longitudinal, one arm, prospective phase II study, designed to evaluate the efficacy of Olanzapine Netupitant and Palonosetron in the controll of nausea and vomiting induced by highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
The population of the study is women diagnosed with breast cancer, who will start chemotherapy (Doxorubicine and Cyclophosfamide). We will evaluate the control of nausea and vomiting in the first cycle of chemotherapy, utilizing Netupitant (300mg) + palonosetron (0,56mg) in day 1 and Olanzapine 5mg starting on Day 0, given once a day for five days. The primary endpoint of this study is complete response rate (no nausea, no emesis no use of rescue medication).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer hitologically confirmed
* 18 Years and older (Adult, Older Adult)
* Patients about to start use of Doxorubicine 60mg/m2 + Cyclophosfamide 600mg/m2
* No previous chemotherapy for breast cancer

Exclusion Criteria:

* Patients not capable of completing the questionnaire
* Patients with other condition that could cause nausea and emesis
* Use of opioids
* Use of antipsychotic medications
* Patients not capable of taking medications orally

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Nausea Complete Response Rate | 5 days after chemotherapeutic administration
  Defined as no nausea and no rescue medication

SECONDARY OUTCOMES:
Complete Emesis Control | For the following time periods: 0-24 hours (acute), 24+ to 120 hours (delayed), and 0-120 hours (overall)
  Defined as no emetic episodes and no use of rescue medications
Complete Control | For the following time periods: 0-24 hours (acute), 24+ to 120 hours (delayed), and 0-120 hours (overall)
  Defined as no nausea, no emesis and no rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Rebouças, MD, Principal Investigator — Instituto Brasileiro de Controle do Cancer
Locations (1):
- IBCC Oncologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Razvi Y, Chan S, McFarlane T, McKenzie E, Zaki P, DeAngelis C, Pidduck W, Bushehri A, Chow E, Jerzak KJ. ASCO, NCCN, MASCC/ESMO: a comparison of antiemetic guidelines for the treatment of chemotherapy-induced nausea and vomiting in adult patients. Support Care Cancer. 2019 Jan;27(1):87-95. doi: 10.1007/s00520-018-4464-y. Epub 2018 Oct 3. PMID 30284039
- [Background] Roila F, Molassiotis A, Herrstedt J, Aapro M, Gralla RJ, Bruera E, Clark-Snow RA, Dupuis LL, Einhorn LH, Feyer P, Hesketh PJ, Jordan K, Olver I, Rapoport BL, Roscoe J, Ruhlmann CH, Walsh D, Warr D, van der Wetering M; participants of the MASCC/ESMO Consensus Conference Copenhagen 2015. 2016 MASCC and ESMO guideline update for the prevention of chemotherapy- and radiotherapy-induced nausea and vomiting and of nausea and vomiting in advanced cancer patients. Ann Oncol. 2016 Sep;27(suppl 5):v119-v133. doi: 10.1093/annonc/mdw270. No abstract available. PMID 27664248
- [Background] Gralla R, Lichinitser M, Van Der Vegt S, Sleeboom H, Mezger J, Peschel C, Tonini G, Labianca R, Macciocchi A, Aapro M. Palonosetron improves prevention of chemotherapy-induced nausea and vomiting following moderately emetogenic chemotherapy: results of a double-blind randomized phase III trial comparing single doses of palonosetron with ondansetron. Ann Oncol. 2003 Oct;14(10):1570-7. doi: 10.1093/annonc/mdg417. PMID 14504060
- [Background] Wang H, Wang Y, Rayburn ER, Hill DL, Rinehart JJ, Zhang R. Dexamethasone as a chemosensitizer for breast cancer chemotherapy: potentiation of the antitumor activity of adriamycin, modulation of cytokine expression, and pharmacokinetics. Int J Oncol. 2007 Apr;30(4):947-53. PMID 17332934
- [Background] Kim MH, Kim DW, Park S, Kim JH, Lee KY, Hwang J, Yoo YC. Single dose of dexamethasone is not associated with postoperative recurrence and mortality in breast cancer patients: a propensity-matched cohort study. BMC Cancer. 2019 Mar 20;19(1):251. doi: 10.1186/s12885-019-5451-5. PMID 30894164
- [Background] Chen YX, Wang Y, Fu CC, Diao F, Song LN, Li ZB, Yang R, Lu J. Dexamethasone enhances cell resistance to chemotherapy by increasing adhesion to extracellular matrix in human ovarian cancer cells. Endocr Relat Cancer. 2010 Jan 29;17(1):39-50. doi: 10.1677/ERC-08-0296. Print 2010 Mar. PMID 19776289
- [Background] Obradovic MMS, Hamelin B, Manevski N, Couto JP, Sethi A, Coissieux MM, Munst S, Okamoto R, Kohler H, Schmidt A, Bentires-Alj M. Glucocorticoids promote breast cancer metastasis. Nature. 2019 Mar;567(7749):540-544. doi: 10.1038/s41586-019-1019-4. Epub 2019 Mar 13. PMID 30867597
- [Background] de Castro Baccarin AL, Irene MN, de Iracema Gomes Cubero D, Luz AS, Castro SN, Sordi R, Moz LES, Del Giglio A. The feasibility of dexamethasone omission in weekly paclitaxel treatment for breast cancer patients. Support Care Cancer. 2019 Mar;27(3):927-931. doi: 10.1007/s00520-018-4381-0. Epub 2018 Aug 1. PMID 30069696
- [Background] Navari RM, Nagy CK, Gray SE. The use of olanzapine versus metoclopramide for the treatment of breakthrough chemotherapy-induced nausea and vomiting in patients receiving highly emetogenic chemotherapy. Support Care Cancer. 2013 Jun;21(6):1655-63. doi: 10.1007/s00520-012-1710-6. Epub 2013 Jan 12. PMID 23314603
- [Background] Cruz FM, de Iracema Gomes Cubero D, Taranto P, Lerner T, Lera AT, da Costa Miranda M, da Cunha Vieira M, de Souza Fede AB, Schindler F, Carrasco MM, de Afonseca SO, Pinczowski H, del Giglio A. Gabapentin for the prevention of chemotherapy- induced nausea and vomiting: a pilot study. Support Care Cancer. 2012 Mar;20(3):601-6. doi: 10.1007/s00520-011-1138-4. Epub 2011 Apr 5. PMID 21465325
- [Derived] Reboucas CV, Alves RB, Yamada AMTD, Del Giglio A, Cruz FJSM. Omission of dexamethasone in prophylaxis for highly emetogenic chemotherapy in patients with breast cancer. Einstein (Sao Paulo). 2025 May 12;23:eAO1124. doi: 10.31744/einstein_journal/2025AO1124. eCollection 2025. PMID 40367007